CLINICAL TRIAL: NCT01569789
Title: Effects of Auricular Vagus Nerve Stimulation on the Pro-inflammatory Cytokine Response in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Vagus-1
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Cytokine Response to Vagus Nerve Stimulation
Keywords: cytokines; inflammation; vagus nerve; TNF
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ear Stimulation (Active Comparator): Comparing cytokine levels pre and post stimulation of the nerve in the ear
  Interventions: Device: Vagus Nerve Stimulator
- Calf Stimulation (Placebo Comparator): Comparing cytokine levels pre and post stimulation of the placebo area on the calf
  Interventions: Device: Vagus Nerve Stimulator

INTERVENTIONS:
Device: Vagus Nerve Stimulator — Voltage 2, placed on cymba concha
  Arms: Ear Stimulation
Device: Vagus Nerve Stimulator — Voltage 2, place on the placebo area of the calf
  Arms: Calf Stimulation

SUMMARY:
The autonomic (self-regulating) nervous system is important for the function of many organs in the body. The vagus nerve is part of the autonomic nervous system. The vagus nerve carries incoming information from the nervous system to the brain, providing information about what the body is doing, and it also transmits outgoing information which governs a range of reflex responses. It plays an important role in the immune system. A part of the vagus nerve is reachable for stimulation at specific locations in the ear.

The purpose of this study is to better understand how different ways of stimulating the vagus nerve at the ear can affect a chemical marker of inflammation found in human blood that is associated with a variety of inflammatory diseases such as rheumatoid arthritis and lupus. This information may lead to in future studies to see if stimulation of the vagus nerve can improve inflammation in chronic inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years old
* Currently healthy with no medical problems
* Non-smoker

Exclusion Criteria:

* History of any of the following: cardiac arrhythmia, coronary artery disease, chronic inflammatory disease, anemia, malignancy, depression, connective tissue disease (arthritis, vasculitis), neurologic disease, diabetes mellitus, renal disease, malignancy, dementia, psychiatric illness including active psychosis, or any other chronic medical condition
* Use of cholinergic, anti-cholinergic, or beta-blocking medications
* Family history of inflammatory disease
* Pregnancy
* Smoking
* Ear infection (otitis media or externa)
* Implanted vagus nerve stimulator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
TNF levels in the ex vivo LPS-stimulated whole blood | 30 minutes (or 5 days) post stimulation

SECONDARY OUTCOMES:
IL-1B, IL-6, IL-8 and IL-10 levels will also be determined by using the same assay | 30 minutes (or 5 days) post stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Tracey, MD, Principal Investigator — Northwell Health
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

REFERENCES:
- [Derived] Addorisio ME, Imperato GH, de Vos AF, Forti S, Goldstein RS, Pavlov VA, van der Poll T, Yang H, Diamond B, Tracey KJ, Chavan SS. Investigational treatment of rheumatoid arthritis with a vibrotactile device applied to the external ear. Bioelectron Med. 2019 Apr 17;5:4. doi: 10.1186/s42234-019-0020-4. eCollection 2019. PMID 32232095